CLINICAL TRIAL: NCT00155870
Title: Health-Related Quality of Life Among Women Receiving Hysterectomy in National Taiwan University Hospital
Brief Title: Health-Related QoL Among Women Receiving Hysterectomy in NTUH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9200201773
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-12-20 (Estimated); Status verified 2005-06

CONDITIONS: Leiomyoma; Adenomyosis
Keywords: laparoscopic assisted vaginal hysterectomy leiomyoma; adenomyosis; quality of life
MeSH Terms: conditions — Leiomyoma; Adenomyosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: questionnaires

SUMMARY:
Laparoscopic assisted vaginal hysterectomy (LAVH)has become the most prevalent operation method in woman suffering from uterine myoma or adenomyosis nowadays. The operation decisions for these women are always due to symptoms such as pain, anemia and mass effect. However, there is a lack of measurement for these symptoms and therefore highlight the need to validate these symptom by health-related quality of life (QOL) assessments. Patients usually recovered better by LAVH comparing to traditional open surgeries. However, LAVH was restricted to cases with small size uteri and most QOL reported neglected uterine weight or were based on small uteri size. We recently intervened a new surgical procedure called RULU during LAVH and thus released this limitation. This will give a more unbiased study on the effect of QOL in patients receiving LAVH. In this study, we plan to use two questionnaires: the disease specific UFS-QOL and the WHO-QOL Taiwan version questionnaires for patients receiving LAVH. Assessment will be performed before operation; and 3 days, 7 days, 3 months and 18 months after operation. From these assessments, we plan to determine which QOL variables will be useful as operation guidelines for patients suffering from leiomyoma or adenomyosis, and for the assessment of appropriates and outcomes of LAVH.

DETAILED DESCRIPTION:
Hysterectomy is the most common non-pregnancy-related surgical procedure performed in women in Taiwan. There are three surgical approaches to hysterectomy: abdominal, vaginal and laparoscopic assisted vaginal hysterectomy (LAVH) and LAVH has become the most prevalent operation method in woman suffering from uterine myoma or adenomyosis nowadays. The operation decisions for these women are always due to symptoms such as pain, anemia and mass effect. However, there is a lack of measurement for these symptoms and therefore highlight the need to validate these symptom by health-related quality of life (QOL) assessments. Patients usually recovered better by LAVH comparing to traditional open surgeries. However, LAVH was restricted to cases with small size uteri and most QOL reported neglected uterine weight or were based on small uteri size. We recently intervened a new surgical procedure called RULU during LAVH and thus released this limitation. This will give a more unbiased study on the effect of QOL in patients receiving LAVH. In this study, we plan to use two questionnaires: the disease specific UFS-QOL and the WHO-QOL Taiwan version questionnaires for patients receiving LAVH. Assessment will be performed before operation; and 3 days, 7 days, 3 months and 18 months after operation. From these assessments, we plan to determine which QOL variables will be useful as operation guidelines for patients suffering from leiomyoma or adenomyosis, and for the assessment of appropriates and outcomes of LAVH.

ELIGIBILITY:
Inclusion Criteria:

laparoscopic assisted vaginal hysterectomy leiomyoma adenomyosis-

Exclusion Criteria:

other types of operations other types of gynecological disease-

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2005-06; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Torng Pao-Ling, MD, PhD, Principal Investigator — Department of Obstetric and Gynecology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan